CLINICAL TRIAL: NCT07382778
Title: A Multi-center, Open-label, Observational Study to Compare and Evaluate the Efficacy and Safety of Livalozet® According to the Presence or Absence of Diabetes Mellitus in Hypercholesterolemia Patients
Brief Title: Efficacy and Safety of Livalozet® in Hypercholesterolemic Patients With and Without Diabetes
Acronym: VICTORY
Status: Completed | Type: Observational
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: JW21403
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; Diabetes Mellitus; Low Density Lipoprotein Cholesterol; Lipid Profile; Observational Study
MeSH Terms: conditions — Hypercholesterolemia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hypercholesterolemia with Diabetes Mellitus: Observational study; LDL-C and lipid parameters will be followed; no intervention assigned.
- Hypercholesterolemia without Diabetes Mellitus: Observational study; LDL-C and lipid parameters will be followed; no intervention assigned.

SUMMARY:
A Multi-center, Open-label, Observational Study to Compare and Evaluate the Efficacy and Safety of Livalozet® according to the Presence or Absence of Diabetes Mellitus in Hypercholesterolemia Patients

DETAILED DESCRIPTION:
A Multi-center, Open-label, Observational Study

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥19 years
* Diagnosed with hypercholesterolemia
* LDL-C level meets cardiovascular/cerebrovascular risk group classification
* Willing to participate for 12 months
* Provided written informed consent

Exclusion Criteria:

- Contraindications to Livalozet®

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from adult patients aged 19 years or older diagnosed with hypercholesterolemia who are receiving routine clinical care at participating centers. The population includes both patients with and without diabetes mellitus, reflecting real-world treatment practices. Eligible patients must provide informed consent to participate in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 1538 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in LDL-C level at Week 24 | From enrollment to the end of treatment at 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No